CLINICAL TRIAL: NCT02997904
Title: A Randomized Sham Controlled Double Blinded Single Site Clinical Trial Evaluating the Efficacy of Resultz Lice and Egg Elimination Kit for the Removal of Human Head Lice and Eggs on Pediatric and Adult Subjects
Brief Title: A Clinical Trial Evaluating the Efficacy of Resultz Lice and Egg Elimination Kit on Pediatric and Adult Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Piedmont Pharmaceuticals, LLC (Industry)
Collaborators: Lice Solutions Resource Network (LSRN) Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PP-16-001
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-07

CONDITIONS: Pediculus Capitis
Keywords: lice comb; human head lice infestations; combing solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Resultz Lice and Egg Elimination Kit (Experimental): Resultz combing solution, head lice comb and instructions for use in a kit: apply liquid then comb out for 1 hour
  Interventions: Device: Apply Liquid Then Comb Out
- Placebo Lice and Egg Elimination Kit (Placebo Comparator): 20% glycerin combing solution, comb and instructions for use in a kit: apply liquid then comb out for 1 hour
  Interventions: Device: Apply Liquid Then Comb Out

INTERVENTIONS:
Device: Apply Liquid Then Comb Out — Apply liquid to dry hair, wait for 5 minutes, then comb out lice and eggs for up to one hour
  Other Names: Resultz Application

SUMMARY:
A one day study to demonstrate that Resultz Lice and Egg Elimination Kit is statistically superior to a sham control with one hour of combing.

DETAILED DESCRIPTION:
Resultz Lice and Egg Elimination Kit will be efficacious in the removal of human head lice infestations in children and adult subjects under simulated real world conditions.

ELIGIBILITY:
Inclusion Criteria:

* Must have active head lice infestations (at least 1 live louse and eggs)
* Good general health based on medical history
* Each subject has to be consented

Exclusion Criteria:

* Subjects with any condition that would compromise the study
* History of irritation or sensitivity to pediculicides or hair care products
* Subjects with cranial or facial implants
* Subjects who have received radiation within the last 6 months
* Subjects with history of heart disease
* Subjects with history of epilepsy or seizure disorders
* Subjects with neuro-stimulator or pacemaker
* Subject with hair that staff cannot comb
* Subject previously treated in study in last 30 days
* Use of lice treatment in past 2 weeks
* Subject unable to sense pain
* Subject unable to communicate pain

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Shepherd, Principal Investigator — Lice Solutions Resource Network Research
Locations (1):
- Lice Solution Resource Network Research, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Resultz Lice and Egg Removal Kit: Resultz combing solution, head lice comb and instructions for use in a kit: kit used once and combed out for 1 hour
  Resultz Lice and Egg Removal Kit: Clear combing solution, nude colored comb
- Sham Lice and Egg Removal Kit: 20% glycerin combing solution, comb and instructions for use in a kit: kit used once and combed out for 1 hour
  Resultz Lice and Egg Removal Kit: Clear combing solution, nude colored comb
Period: Overall Study
Arm/Group | Resultz Lice and Egg Removal Kit | Sham Lice and Egg Removal Kit
Started | 51 | 49
Completed | 51 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resultz Lice and Egg Removal Kit | Sham Lice and Egg Removal Kit | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.3 (13.5) | 17.8 (12.1) | 16.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 44 | 81
  Male | 14 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 37 | 77
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 49 | 100

OUTCOME MEASURES:

1. Primary Outcome: The Total Number of Lice + Eggs Removed From the Head After One Hour of Combing
Description: A superiority analysis comparing the total number of lice + eggs removed from the head after one hour of combing with the Resultz Kit versus the control. The Resultz Kit was considered a success if the Resultz Kit was superior to the control.
Time Frame: 1 hour
Population: Intent To Treat; including all subjects who were enrolled in the study.
Measure: Mean (Standard Deviation); unit: number of lice and eggs removed
Groups:
- Resultz Lice and Egg Elimination Kit: Resultz combing solution, head lice comb and instructions for use in a kit: kit used once and combed out for 1 hour
  Resultz Lice and Egg Removal Kit: Clear combing solution, nude colored comb
- Sham Lice and Egg Elimination Kit: 20% glycerin combing solution, comb and instructions for use in a kit: kit used once and combed out for 1 hour
  Resultz Lice and Egg Removal Kit: Clear combing solution, nude colored comb
Arm/Group | Resultz Lice and Egg Elimination Kit | Sham Lice and Egg Elimination Kit
Number analyzed (Participants) | 51 | 49
number of lice and eggs removed | 71.3 (61.2) | 26.1 (25.6)
Statistical Analysis 1: Comparison: Resultz Lice and Egg Elimination Kit vs Sham Lice and Egg Elimination Kit; Ho: Total Number of lice and eggs removed with Resultz® ≤ Total number of lice and eggs removed with sham control Ha: Total Number of lice and eggs removed with Resultz® > Total Number of lice and eggs removed with sham control; Test type: Superiority; p < 0.0001, ANOVA; Least Squares Mean Difference = 1.0058, 95% CI 2-sided [0.5829 to 1.4288], Standard Error of Mean 0.2131

2. Secondary Outcome: Total Number of Lice Removed, Total Number of Eggs Removed
Description: Total number of lice removed after one hour of combing and total number of eggs removed after one hour of combing, analyzed separately
Time Frame: 1 hour
Population: Intent To Treat; including all subjects enrolled
Measure: Mean (Standard Deviation); unit: Number of Lice or Number of Eggs
Groups:
- Number or Lice Removed by Resultz: Total number of lice removed after one hour of combing with Resultz; analyzed separately
- Number of Lice Removed by Control: Total number of lice removed after one hour of combing by control; analyzed separately
- Number of Eggs Removed by Resultz: Total number of eggs removed after one hour of combing, analyzed separately
- Number of Eggs Removed by Control: Total number of eggs removed after one hour of combing by control, analyzed separately
Arm/Group | Number or Lice Removed by Resultz | Number of Lice Removed by Control | Number of Eggs Removed by Resultz | Number of Eggs Removed by Control
Number analyzed (Participants) | 51 | 49 | 51 | 49
Number of Lice or Number of Eggs | 40.3 (43.6) | 12 (15.1) | 31 (22.3) | 14.1 (11.8)
Statistical Analysis 1: Comparison: Number or Lice Removed by Resultz vs Number of Lice Removed by Control; Comparison of total number of lice removed and total number of eggs removed were analyzed separately; Test type: Superiority; p < 0.0001, GLIMMX — The P-Values were <0.0001 in both comparison groups; total number lice removed and total number of eggs removed; Least Squares Mean Difference = 1.2084, 95% CI 2-sided [1.1157 to 1.3011], Standard Error of Mean 0.04670
Statistical Analysis 2: Comparison: Number of Eggs Removed by Resultz vs Number of Eggs Removed by Control; Test type: Superiority; p < 0.0001, GLIMMX; Least Squares Mean Difference = 0.7899, 95% CI 2-sided [0.6993 to 0.8805], Standard Error of Mean 0.04565

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Resultz Lice and Egg Removal Kit | Sham Lice and Egg Removal Kit
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 0/51 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not without sponsor permission